CLINICAL TRIAL: NCT04499612
Title: Assessment of the Hemostatic System, Thromboembolic Complications and Cardiovascular Events in Patients With Cardiovascular Implantable Electronic Devices
Brief Title: Influence of Cardiac Implantable Electronic Devices on the Hemostatic System
Status: Completed | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 05/290120
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-10

CONDITIONS: Thromboembolism; Cardiac Event; Hemostatic Disorder
Keywords: Cardiac implantable electronic devices; Pacing; Hemostasis; Thromboembolism; Cardiovascular events; Arrhythmias; Atrial fibrillation; Chronic heart failure
MeSH Terms: conditions — Thromboembolism; Cardiovascular Diseases; Hemostatic Disorders; Arrhythmias, Cardiac; Atrial Fibrillation | interventions — Ultrasonography, Doppler, Duplex; Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group "Single-chamber CIED" (A1): 50 patients with permanent atrial fibrillation and indications for cardiac implantable electronic device implantation (single-chamber system).
  Interventions: Procedure: Cardiac implantable electronic device implantation.; Diagnostic Test: Duplex ultrasound.; Diagnostic Test: Echocardiography.; Diagnostic Test: Blood sampling.
- Group "Dual-chamber CIED" (A2): 50 patients with atrioventricular block/sick sinus syndrome and indications for cardiac implantable electronic device implantation (dual-chamber system).
  Interventions: Procedure: Cardiac implantable electronic device implantation.; Diagnostic Test: Duplex ultrasound.; Diagnostic Test: Echocardiography.; Diagnostic Test: Blood sampling.
- Group "Dual-chamber CIED + Atrial fibrillation" (A3): 50 patients with atrioventricular block/sick sinus syndrome, paroxysmal or persistent atrial fibrillation and indications for cardiac implantable electronic device implantation (dual-chamber system).
  Interventions: Procedure: Cardiac implantable electronic device implantation.; Diagnostic Test: Duplex ultrasound.; Diagnostic Test: Echocardiography.; Diagnostic Test: Blood sampling.
- Group "CIED Replace" (B): 50 patients with cardiac implantable electronic device implantation 6-12 years ago (single- or dual-chamber system).
  Interventions: Procedure: Cardiac implantable electronic device replace.; Diagnostic Test: Duplex ultrasound.; Diagnostic Test: Echocardiography.; Diagnostic Test: Blood sampling.
- Group "Conservative" (C): 50 patients with atrioventricular block/sick sinus syndrome/atrial fibrillation and without indications for cardiac implantable electronic device implantation (conservative group).
  Interventions: Diagnostic Test: Duplex ultrasound.; Diagnostic Test: Echocardiography.; Diagnostic Test: Blood sampling.

INTERVENTIONS:
Procedure: Cardiac implantable electronic device implantation. — Patients who have indications will receive cardiac implantable electronic device implantation.
  Groups: Group "Dual-chamber CIED + Atrial fibrillation" (A3); Group "Dual-chamber CIED" (A2); Group "Single-chamber CIED" (A1)
Procedure: Cardiac implantable electronic device replace. — Patients who have indications will receive cardiac implantable electronic device replace.
  Groups: Group "CIED Replace" (B)
Diagnostic Test: Duplex ultrasound. — Patients will undergo ultrasound examination of the vessels of the upper and lower extremities.
Diagnostic Test: Echocardiography. — Patients will undergo an ultrasound examination of the heart.
Diagnostic Test: Blood sampling. — Patients will be taken venous blood to determine the studied markers of hemostasis system.

SUMMARY:
The hemostasis system is one of the many biological systems of the human body, designed to preserve the liquid state of blood and prevent its loss during vascular injuries. The ideal balance between its coagulant and anticoagulant components never occurs. In various diseases and pathological conditions, the balance of the hemostasis system may be disturbed. Shifts towards hypercoagulability lead to the development of hemorrhagic complications, opposite shifts lead to the development of thrombotic complications.

Patients with cardiac implantable electronic devices (CIED) are not rare and unique, today doctors meet with them every day. Its more than 1.5 million CIED's implanted every year.

Before surgery these patients are standard cardiology department patients with chronic heart failure (CHF), which develops due to the presence of arrhythmias, coronary heart disease, hypertension, congenital heart disease, myocardial infarction, myocarditis or other diseases and conditions. CHF is the most common, severe and unfavorable prognostic complication of these diseases. With CHF, the balance of the hemostasis system shifts towards hypercoagulation. Patients with CHF have an increased risk of arterial and venous thrombosis, pulmonary embolism, myocardial infarction, stroke, numerous brady- and tachyarrhythmias and other complications.

After CIED implantation, bradyarrhythmia is eliminated, as one of the parts in the pathogenesis of CHF. Patients, especially those with severe symptoms, improve their condition in the early postoperative period. In the long-term period, pacing, on the contrary, may contribute to the progression of CHF. The wrong choice of pacing mode or the place of electrode implantation can lead to desynchronization of the heart chambers, myocardial remodeling and left ventricular dysfunction.

Uncertainty is also observed in relation to the hemostasis system after CIED implantation. On the one hand, correction of bradyarrhythmia and CHF should provide patients with a shift towards hypocoagulability by normalizing the heart rate. On the other hand, trauma to the vessel wall during surgery, further placement of the CIED leads in the vessels, and perioperative stress can lead to even greater shifts towards hypercoagulation.

DETAILED DESCRIPTION:
250 patients of similar age, gender, and ethnicity will be divided into five groups: Group A1-3: 150 patients with indications for cardiac implantable electronic device (CIED) implantation; Group B: 50 patients with an CIED implanted 8-10 years ago; Group C: 50 patients with diseases similar to group A, but without indications for CIED implantation; Patients will be followed up for 2 years. Patients of group A1-3 will be taken peripheral venous blood to assess the studied parameters of hemostasis (platelet count, plateletcrit, mean platelet volume, platelet distribution width, von Willebrand factor, P-selectin, coagulation factor I (FI), coagulation factor II (FII), coagulation factor V (FV), coagulation factor VII (FVII), coagulation factor X (FX), coagulation factor VIII (FVIII), coagulation factor IX (FIX), coagulation factor XI (FXI), coagulation factor XII (FXII), plasminogen, soluble fibrin, plasminogen activator inhibitor-1 (PAI-1), D-dimer, antithrombin III, protein C) and duplex ultrasound of the vessels of the upper and lower extremities before the operation, after 7 days, 1 and 12 months after the operation. Similar procedures will be performed for patients of groups B and C only when included in the study. Echocardiography will be performed on all patients at enrollment, after 12 and 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* for group A1-3: atrioventricular block/sick sinus syndrome/atrial fibrillation with impaired conduction as indications for cardiac implantable electronic device implantation;
* for group B: atrioventricular block/sick sinus syndrome/atrial fibrillation with impaired conduction and cardiac implantable electronic device implanted 6-12 years ago;
* for group C: atrioventricular block/sick sinus syndrome/atrial fibrillation with impaired conduction without indications for cardiac implantable electronic device implantation.

Exclusion Criteria:

* active cancer or a remission period of less than 5 years;
* decompensated somatic pathology;
* pregnancy or breastfeeding in women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment in cardiology and cardiac surgery departments who have an implanted cardiac implantable electronic device or have indication/no indication for cardiac implantable electronic device implantation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Development of thromboembolism: venous thrombosis, pulmonary embolism, arterial thrombosis, arterial thromboembolism, transient ischemic attack, stroke. | Up to 2 years after enrollment (according to the study design).
  Development of thromboembolic complications after the cardiac implantable electronic device implantation/replace or thromboembolism in conservative group patients during observation period.
Development of cardiovascular event: myocardial infarction, acute coronary syndrome, atrial fibrillation, decompensation of chronic heart failure. | Up to 2 years after enrollment (according to the study design).
  Development of cardiovascular events after the cardiac implantable electronic device implantation/replace or in conservative group patients during observation period.

SECONDARY OUTCOMES:
Hemostasis system markers deviations. | Up to 2 years after enrollment (according to the study design).
  Deviation of investigated markers of the hemostasis system from normal values.

CONTACTS AND LOCATIONS:
Overall Officials: Igor A. Suchkov, MD, DSc, Principal Investigator — Ryazan State Medical University
Locations (1):
- Ryazan State Medical University, Ryazan, Ryazan Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Basic demographic data, including sex, age, and ethnicity are to be shared if allowed by the privacy policy.

REFERENCES:
- [Background] Kalinin RE, Suchkov IA, Shitov II, Mzhavanadze ND, Povarov VO. [Venous thromboembolic complications in patients with cardiovascular implantable electronic devices]. Angiol Sosud Khir. 2017;23(4):69-74. Russian. PMID 29240058